CLINICAL TRIAL: NCT06750406
Title: Effects of Mind Body Exercises on Stress, Anxiety and Fatigue in Pregnant Women
Brief Title: Effects of Mind Body Exercises in Pregnant Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REC/RCR&AHS/24/0529
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy Related
Keywords: pregnant women; exercises; yoga; anxiety; fatigue
MeSH Terms: conditions — Motor Activity; Anxiety Disorders; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mind body exercises (Experimental): The intervention consists of a structured program of mind-body exercises designed specifically for pregnant women. This involves a combination of yoga sessions, mindfulness meditation practices, deep breathing exercises, and progressive muscle relaxation techniques. The duration of these sessions will be 45 to 60 minutes each, with a recommended frequency of 2-3 times per week for eight weeks
  Interventions: Other: mind body exercises
- Relaxation exercises (Active Comparator): this includes Awareness about relaxation exercises including relax postures and generalized exercise interventions. The duration of these sessions will be 45 to 60 minutes each, with a recommended frequency of 2-3 times per week for eight weeks
  Interventions: Other: relaxation exercises

INTERVENTIONS:
Other: mind body exercises — intervention might consist of a structured program of mind-body exercises designed specifically for pregnant women. This could involve a combination of yoga sessions, mindfulness meditation practices, deep breathing exercises, and progressive muscle relaxation techniques. The duration of these sessions will be 45 to 60 minutes each, with a recommended frequency of 2-3 times per week for 8 weeks
  Arms: mind body exercises
Other: relaxation exercises — It involves relaxation exercises including deep breathing, relaxing postures etc. The duration of these sessions will be 45 to 60 minutes each, with a recommended frequency of 2-3 times per week for 8 weeks
  Arms: Relaxation exercises

SUMMARY:
his Study is a randomized controlled trial (RCT) which will be collected through non probability convenient sampling technique and will be carried out for 10 months duration with a sample size of 34 pregnant women which will be collected through non probability convenient sampling technique. the participants will be divided into two groups. Group A will be involved in mind body exercises and group B will be given relaxation exercises

DETAILED DESCRIPTION:
This Study is a randomized controlled trial (RCT) which will be collected through non probability convenient sampling technique and will be carried out for 10 months duration with a sample size of 34 pregnant women which will be collected through non probability convenient sampling technique. Sample will be collected from Gosha shifa and Ishaq Haroon Hospital. Pregnant women in their second trimester (between 14-28 weeks). Age between 20 to 35 years. Able to understand and participate in mind-body exercises sessions will be included. High-risk pregnancies (e.g., gestational diabetes, hypertension). Pre-existing medical conditions that could interfere with participation (e.g., severe musculoskeletal disorders). will be excluded. Tools used in the study are perceived stress scale (PSS) , Hamilton Anxiety Rating Scale (HARS) and Fatigue severity scale-(FSS).Data will be analyzed by busing SPSS 26.0

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in their second trimester (between 14-28 weeks)
* Primi gravid
* Able to understand and participate in mind-body exercises sessions

Exclusion Criteria:

* High-risk pregnancies (e.g., gestational diabetes, hypertension)
* Pre-existing medical conditions that could interfere with participation (e.g., severe musculoskeletal disorders)
* History of psychiatric disorders requiring ongoing treatment
* History of miscarriage

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant females
Enrollment: 34 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Perceived- Stress Scale (PSS) | 8th week
  The PSS has shown good internal consistency, with Cronbach's alpha coefficients typically ranging from 0.70 to 0.90. Test-retest reliability over short intervals (e.g., a few days to a month) is generally acceptable, with correlation coefficients often above 0.70.The PSS correlates well with other measures of stress and related constructs, demonstrating good construct validity. High PSS scores have been associated with increased risk for health problems and psychological issues, indicating good predictive validity
Hamilton Anxiety Rating Scale (HARS) | 8th week
  The HARS has demonstrated good internal consistency, with Cronbach's alpha coefficients typically ranging from 0.74 to 0.96. Inter-rater reliability is high, with intraclass correlation coefficients often above 0.80. Test-retest reliability over periods of days to weeks is generally good, with correlation coefficients often above 0.75.The HARS covers a broad range of anxiety symptoms, ensuring good content validity. It correlates well with other measures of anxiety and related constructs, demonstrating good construct validity. The HARS scores are consistent with clinical diagnoses of anxiety disorders, indicating good concurrent validity
Fatigue Severity Scale (FSS) | 8th week
  The FSS has shown excellent internal consistency, with Cronbach's alpha coefficients typically above 0.90. Test-retest reliability over periods ranging from a few days to several weeks is generally high, with correlation coefficients often above 0.80.The FSS includes items that comprehensively cover the domain of fatigue, ensuring good content validity. It correlates well with other measures of fatigue and related constructs, demonstrating good construct validity. The FSS scores are consistent with clinical assessments of fatigue severity, indicating good concurrent validity

CONTACTS AND LOCATIONS:
Overall Officials: hina gul, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Ishaq Haroon hospital and Goshea shifa hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng YC, Su MI, Liu CW, Huang YC, Huang WL. Heart rate variability in patients with anxiety disorders: A systematic review and meta-analysis. Psychiatry Clin Neurosci. 2022 Jul;76(7):292-302. doi: 10.1111/pcn.13356. Epub 2022 Apr 27. PMID 35340102
- [Background] Evans K, Spiby H, Morrell JC. Non-pharmacological interventions to reduce the symptoms of mild to moderate anxiety in pregnant women. A systematic review and narrative synthesis of women's views on the acceptability of and satisfaction with interventions. Arch Womens Ment Health. 2020 Feb;23(1):11-28. doi: 10.1007/s00737-018-0936-9. Epub 2019 Jan 7. PMID 30613846
- [Background] Traylor CS, Johnson JD, Kimmel MC, Manuck TA. Effects of psychological stress on adverse pregnancy outcomes and nonpharmacologic approaches for reduction: an expert review. Am J Obstet Gynecol MFM. 2020 Nov;2(4):100229. doi: 10.1016/j.ajogmf.2020.100229. Epub 2020 Sep 24. PMID 32995736
- [Background] Nadholta P, Kumar K, Saha PK, Suri V, Singh A, Anand A. Mind-body practice as a primer to maintain psychological health among pregnant women-YOGESTA-a randomized controlled trial. Front Public Health. 2023 Sep 12;11:1201371. doi: 10.3389/fpubh.2023.1201371. eCollection 2023. PMID 37766749
- [Background] Oyarzabal I, Zabala-Lekuona A, Mota AJ, Palacios MA, Rodriguez-Dieguez A, Lorusso G, Evangelisti M, Rodriguez-Esteban C, Brechin EK, Seco JM, Colacio E. Magneto-thermal properties and slow magnetic relaxation in Mn(II)Ln(III) complexes: influence of magnetic coupling on the magneto-caloric effect. Dalton Trans. 2022 Aug 30;51(34):12954-12967. doi: 10.1039/d2dt01869a. PMID 35960153
- [Background] Guo P, Zhang X, Liu N, Wang J, Chen D, Sun W, Li P, Zhang W. Mind-body interventions on stress management in pregnant women: A systematic review and meta-analysis of randomized controlled trials. J Adv Nurs. 2021 Jan;77(1):125-146. doi: 10.1111/jan.14588. Epub 2020 Oct 13. PMID 33048358
- [Background] Lerdal A. Fatigue severity scale. Encyclopedia of quality of life and well-being research: Springer; 2021. p. 1-5.